CLINICAL TRIAL: NCT05497700
Title: Comparison of Ephedrine Versus Norepinephrine Efficacity to Correct Anesthesia Induction Related Hypotension in Chronic Renal Insufficiency Patients
Brief Title: Comparative Efficacity of Ephedrine Versus Norepinephrine to Correct Anesthesia Induction Related Hypotension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, department of Anesthesiology, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VASO_IRC
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Hypotension on Induction
MeSH Terms: interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drug will be prepared by an anesthesia nurse not involved in the care of the patient and labeled as "VASO-IRC-inclusion number".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ephedrine group (Active Comparator): In this group, any hypotension less than 65 mm Hg will be corrected by bolus injection of 6 mg ephedrine. Bolus injection will be repeated every 3 minutes, as needed, to keep mean arterial pressure above 65 mm Hg.
  Interventions: Drug: Ephedrine
- Norepinephrine group (Experimental): In this group, any hypotension less than 65 mm Hg will be corrected by bolus injection of 6 mcg norepinephrine. Bolus injection will be repeated every 3 minutes, as needed, to keep mean arterial pressure above 65 mm Hg.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Ephedrine — Bolus injection of 6 mg ephedrine to keep mean arterial blood pressure above 65 mm Hg
  Arms: Ephedrine group
Drug: Norepinephrine — Bolus injection of either 6 mcg norepinephrine to keep mean arterial blood pressure above 65 mm Hg
  Arms: Norepinephrine group

SUMMARY:
Hypotension occurs frequently after anesthesia induction and is more frequent in patients with chronic renal insufficiency. This hypotension occurs most frequently during the 20 minutes after anesthesia induction. Hypotension is commonly corrected by ephedrine bolus injection. However, presynaptic noradrenaline reserve may be lower in patients with chronic renal insufficiency rendering this treatment less effective. Another drug commonly used is norepinephrine, which action is independent of presynaptic noradrenaline storage.

The primary hypothesis is that in patients with chronic renal insufficiency, bolus injection of norepinephrine will be more effective then ephedrine injections to correct hypotension after anesthesia induction.

60 patients with a glomerular filtration rate less than 45 mL/min/m2 (KDIGO classification less than grade 3b) will be included in this prospective double blind trial. All patients will be anesthetized by target-controlled infusion of propofol adjusted to a patient state index (Measured by Sedline, Masimo) of 25-50. Sufentanil injection will be based on noxious stimuli according to the attending anesthesiologist's judgement.

Non-invasive blood pressure will be measured at the pre-anesthesia clinic, before induction and every minute up to 20 minutes post anesthesia induction. Episodes of hypotension, defined as a mean arterial blood pressure less than 65 mm Hg, will be treated either by a bolus injection of 6 mg ephedrine or a bolus injection of 6 mcg norepinephrine, which are equipotent doses. Seringues containing either ephedrine 3 mg/mL or norepinephrine 3 mcg/mL will be prepared by an anesthesia nurse not involved in the care of the patient and labeled as "VASO-IRC-inclusion number". Randomization will be done by a computer generated list in a block randomization of 5.

Primary outcome is the number of boluses needed to maintain arterial blood pressure above a mean of 65 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery
* general anesthesia
* chronic renal insufficiency defined as a glomerular filtration rate < 45 mL/min/m2

Exclusion Criteria:

* cardiac insufficiency with a left ventricular ejection fraction < 50%
* severe cardiomyopathy
* severe cardiac valvular disease
* use of enzyme converting inhibitors or sartans less than 24h before surgery
* use of alpha2 antihypertension medication
* chronic treatment by: noradrenaline or dopamine recapture inhibitors, tricyclic antidepressants, monoamine oxidase inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of boluses | 20 minutes after anesthesia induction
  Primary outcome is the number of boluses of either ephedrine or norepinephrine needed to keep mean arterial blood pressure above 65 mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cockwell P, Fisher LA. The global burden of chronic kidney disease. Lancet. 2020 Feb 29;395(10225):662-664. doi: 10.1016/S0140-6736(19)32977-0. Epub 2020 Feb 13. No abstract available. PMID 32061314
- [Background] Gansevoort RT, Correa-Rotter R, Hemmelgarn BR, Jafar TH, Heerspink HJ, Mann JF, Matsushita K, Wen CP. Chronic kidney disease and cardiovascular risk: epidemiology, mechanisms, and prevention. Lancet. 2013 Jul 27;382(9889):339-52. doi: 10.1016/S0140-6736(13)60595-4. Epub 2013 May 31. PMID 23727170
- [Background] Deng J, Lenart J, Applegate RL. General anesthesia soon after dialysis may increase postoperative hypotension - A pilot study. Heart Lung Vessel. 2014;6(1):52-9. PMID 24800198
- [Background] Schmidt IM, Hubner S, Nadal J, Titze S, Schmid M, Barthlein B, Schlieper G, Dienemann T, Schultheiss UT, Meiselbach H, Kottgen A, Floge J, Busch M, Kreutz R, Kielstein JT, Eckardt KU. Patterns of medication use and the burden of polypharmacy in patients with chronic kidney disease: the German Chronic Kidney Disease study. Clin Kidney J. 2019 May 24;12(5):663-672. doi: 10.1093/ckj/sfz046. eCollection 2019 Oct. PMID 31584562
- [Background] Zoccali C, Mallamaci F, Parlongo S, Cutrupi S, Benedetto FA, Tripepi G, Bonanno G, Rapisarda F, Fatuzzo P, Seminara G, Cataliotti A, Stancanelli B, Malatino LS. Plasma norepinephrine predicts survival and incident cardiovascular events in patients with end-stage renal disease. Circulation. 2002 Mar 19;105(11):1354-9. doi: 10.1161/hc1102.105261. PMID 11901048
- [Background] Grassi G, Quarti-Trevano F, Seravalle G, Arenare F, Volpe M, Furiani S, Dell'Oro R, Mancia G. Early sympathetic activation in the initial clinical stages of chronic renal failure. Hypertension. 2011 Apr;57(4):846-51. doi: 10.1161/HYPERTENSIONAHA.110.164780. Epub 2011 Feb 7. PMID 21300663
- [Background] Converse RL Jr, Jacobsen TN, Toto RD, Jost CM, Cosentino F, Fouad-Tarazi F, Victor RG. Sympathetic overactivity in patients with chronic renal failure. N Engl J Med. 1992 Dec 31;327(27):1912-8. doi: 10.1056/NEJM199212313272704. PMID 1454086
- [Background] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Background] Mathis MR, Naik BI, Freundlich RE, Shanks AM, Heung M, Kim M, Burns ML, Colquhoun DA, Rangrass G, Janda A, Engoren MC, Saager L, Tremper KK, Kheterpal S, Aziz MF, Coffman T, Durieux ME, Levy WJ, Schonberger RB, Soto R, Wilczak J, Berman MF, Berris J, Biggs DA, Coles P, Craft RM, Cummings KC, Ellis TA 2nd, Fleishut PM, Helsten DL, Jameson LC, van Klei WA, Kooij F, LaGorio J, Lins S, Miller SA, Molina S, Nair B, Paganelli WC, Peterson W, Tom S, Wanderer JP, Wedeven C; Multicenter Perioperative Outcomes Group Investigators. Preoperative Risk and the Association between Hypotension and Postoperative Acute Kidney Injury. Anesthesiology. 2020 Mar;132(3):461-475. doi: 10.1097/ALN.0000000000003063. PMID 31794513
- [Background] Camilleri JF, Barragan P, Massonat J, Moyal C, Jouve B, Durand C, Collet F, Gerard R. [Acute occlusion of the renal artery caused by an embolism of cardiac origin. Treatment by in situ thrombolysis]. Arch Mal Coeur Vaiss. 1989 Jul-Aug;82(8):1473-6. French. PMID 2508602
- [Background] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2017 Aug 4;8(8):CD002251. doi: 10.1002/14651858.CD002251.pub3. PMID 28976555
- [Background] Ali Elnabtity AM, Selim MF. Norepinephrine versus Ephedrine to Maintain Arterial Blood Pressure during Spinal Anesthesia for Cesarean Delivery: A Prospective Double-blinded Trial. Anesth Essays Res. 2018 Jan-Mar;12(1):92-97. doi: 10.4103/aer.AER_204_17. PMID 29628561
- [Background] Hassani V, Movaseghi G, Safaeeyan R, Masghati S, Ghorbani Yekta B, Farahmand Rad R. Comparison of Ephedrine vs. Norepinephrine in Treating Anesthesia-Induced Hypotension in Hypertensive Patients: Randomized Double-Blinded Study. Anesth Pain Med. 2018 Aug 26;8(4):e79626. doi: 10.5812/aapm.79626. eCollection 2018 Aug. PMID 30271750
- [Background] Xu S, Mao M, Zhang S, Qian R, Shen X, Shen J, Wang X. A randomized double-blind study comparing prophylactic norepinephrine and ephedrine infusion for preventing maternal spinal hypotension during elective cesarean section under spinal anesthesia: A CONSORT-compliant article. Medicine (Baltimore). 2019 Dec;98(51):e18311. doi: 10.1097/MD.0000000000018311. PMID 31860981
- [Background] Schnider TW, Minto CF, Gambus PL, Andresen C, Goodale DB, Shafer SL, Youngs EJ. The influence of method of administration and covariates on the pharmacokinetics of propofol in adult volunteers. Anesthesiology. 1998 May;88(5):1170-82. doi: 10.1097/00000542-199805000-00006. PMID 9605675
- [Background] Beierwaltes WH, Carretero OA, Scicli AG. Renal hemodynamics in response to a kinin analogue antagonist. Am J Physiol. 1988 Sep;255(3 Pt 2):F408-14. doi: 10.1152/ajprenal.1988.255.3.F408. PMID 3414801
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066